CLINICAL TRIAL: NCT02337062
Title: Randomised, Double-blind, Placebo-controlled Phase III Study of APD421 (Amisulpride for IV Injection) as Combination Prophylaxis Against Post-operative Nausea and Vomiting in High-risk Patients
Brief Title: Phase IIIb Study of APD421 in Combination as PONV Prophylaxis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acacia Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DP10017
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Results first posted 2017-08-04 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: PONV
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- APD421 + standard anti-emetic (Experimental): Single dose of IV APD421
  Interventions: Drug: APD421
- Placebo + standard anti-emetic (Placebo Comparator): Single dose of IV placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APD421
  Arms: APD421 + standard anti-emetic
Drug: Placebo
  Arms: Placebo + standard anti-emetic

SUMMARY:
A comparison of the efficacy of APD421 and placebo when combined with a standard anti-emetic in the prevention of PONV in patients at high risk of Post-operative Nausea and Vomiting (PONV).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* Patients undergoing elective surgery (open or laparoscopic technique) under general anaesthesia, expected to last at least one hour from induction of anaesthesia to wound closure
* Patients with at least 3 "Apfel" risk factors for PONV

Exclusion Criteria:

* Patients scheduled to undergo transplant surgery
* Patients scheduled to receive only a local anaesthetic/regional neuraxial (intrathecal or epidural) block
* Patients who are expected to remain ventilated for a period after surgery
* Patients who are expected to need a naso- or orogastric tube in situ after surgery is completed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1147 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kranke, MD, Principal Investigator — Würzburg University Hospitals
Locations (25):
- United States (14):
  - Helen Keller Hospital, Sheffield, Alabama
  - UCSF School of Medicine, San Francisco, California
  - Jackson Memorial Hospital, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Albany Medical Center Hospital, Albany, New York
  - Stony Brook Medicine, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - First Street Surgical Center, Bellaire, Texas
  - Victory Medical Center Houston, Houston, Texas
  - Memorial Hermann-Memorial City Hospital, Houston, Texas
- France (5):
  - University Hospital, Besançon
  - Centre Hospitalier Lyon-Sud, Lyon
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Hopital Foch, Paris
  - CHU de Hautepierre, Strasbourg
- Germany (6):
  - HELIOS Klinikum Aue, Aue
  - Universitätsklinikum Bonn, Bonn
  - Klinikum Ludwigshafen, Ludwigshafen
  - Universitätsmedizin Mainz, Mainz
  - Philipps University, Marburg
  - University Hospitals of Würzburg, Würzburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study start date:- 12th February 2015 (first patient in)
  Study completion date:- 28th September 2015 (last patient last visit)
  Location:-France, Germany and the USA.
Groups:
- APD421 + Standard Anti-emetic: APD421 (amisulpride) at 5 mg administered as a single, slow, intravenous (IV) push over one minute at the time of induction of anaesthesia; given in combination with standard anti-emetic.
- Placebo + Standard Anti-emetic: Matching Placebo administered as a single, slow push, IV push over one minute at the time of induction anaesthesia given in combination with standard anti-emetic
Period: Overall Study
Arm/Group | APD421 + Standard Anti-emetic | Placebo + Standard Anti-emetic
Started | 572 | 575
Completed | 555 | 556
Not Completed | 17 | 19

BASELINE CHARACTERISTICS:
Groups:
- APD421 + Standard Anti-emetic: Single dose of IV APD421
  APD421
- Placebo + Standard Anti-emetic: Single dose of IV placebo
  Placebo
- Total: Total of all reporting groups
Arm/Group | APD421 + Standard Anti-emetic | Placebo + Standard Anti-emetic | Total
Number analyzed (Participants) | 572 | 575 | 1147
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.8 (14.24) | 48.3 (13.98) | 48.5 (14.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 552 | 557 | 1109
  Male | 20 | 18 | 38
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 353 | 351 | 704
  France | 79 | 85 | 164
  Germany | 140 | 139 | 279

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response
Description: Complete response defined as no emesis and no use of rescue medication in the 24 hour period after end of surgery (defined as wound closure)
Time Frame: 24 hours after the end of surgery
Population: Modified intent-to-treat
Measure: Count of Participants; unit: Participants
Groups:
- APD421 5mg + Standard Anti-emetic: APD421 (amisulpride) at 5 mg administered as a single, slow, intravenous (IV) push over one minute at the time of induction of anaesthesia; given in combination with standard anti-emetic.
- Placebo + Standard Anti-emetic: Matching placebo administered as a single, slow, IV push over one minute, at the time of induction of anaesthesia; given in combination with standard anti-emetic
Arm/Group | APD421 5mg + Standard Anti-emetic | Placebo + Standard Anti-emetic
Number analyzed (Participants) | 572 | 575
Participants | 330 | 268
Statistical Analysis 1: Comparison: APD421 5mg + Standard Anti-emetic vs Placebo + Standard Anti-emetic; The primary efficacy analysis was a comparison of the incidence of the primary efficacy variable between the two groups that received APD421 and the group that received placebo, using Pearson's χ2 test; Test type: Superiority; p < 0.001, Chi-squared — The threshold for determining statistical significance in the comparison of incidence of success between the active and placebo groups (the primary efficacy analysis) was a p-value of 2.5% one-sided

2. Secondary Outcome: Number of Participants With Emesis
Description: Emesis is defined as vomiting (production of even the smallest amount of stomach contents) or retching (muscular movements of vomiting but without expulsion of stomach contents, usually because of an empty stomach)
Time Frame: 24 hours after the end of surgery
Measure: Count of Participants; unit: Participants
Groups:
- APD421 5mg + Standard Anti-emetic: Single IV dose of 5 mg APD421 administered in combination with standard anti-emetic
- Placebo + Standard Anti-emetic: Single dose of IV placebo administered in combination with standard anti-emetic
Arm/Group | APD421 5mg + Standard Anti-emetic | Placebo + Standard Anti-emetic
Number analyzed (Participants) | 572 | 575
Participants | 79 | 115
Statistical Analysis 1: Comparison: APD421 5mg + Standard Anti-emetic vs Placebo + Standard Anti-emetic; Test type: Superiority; p = 0.003, Chi-squared

3. Secondary Outcome: Number of Participants Receiving Rescue Medication
Description: Rescue medication defined as an antiemetic (or other medication) given with the intention of relieving nausea and/or emesis, or any incidental use of a drug known to have antiemetic potential
Time Frame: 24 hours after the end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 5mg + Standard Anti-emetic | Placebo + Standard Anti-emetic
Number analyzed (Participants) | 572 | 575
Participants | 234 | 284
Statistical Analysis 1: Comparison: APD421 5mg + Standard Anti-emetic vs Placebo + Standard Anti-emetic; Test type: Superiority; p = 0.002, Chi-squared

4. Secondary Outcome: Number of Participants With Any Nausea
Description: Nausea (defined as the desire to vomit without the presence of expulsive muscular movements) measured on a 0-10 verbal response scale, where 0=no nausea at all and 10=the worst nausea imaginable. "Any nausea" means a score ≥ 1.
Time Frame: 24 hours after the end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 5mg + Standard Anti-emetic | Placebo + Standard Anti-emetic
Number analyzed (Participants) | 572 | 575
Participants | 286 | 335
Statistical Analysis 1: Comparison: APD421 5mg + Standard Anti-emetic vs Placebo + Standard Anti-emetic; Test type: Superiority; p = 0.002, Chi-squared

5. Secondary Outcome: Number of Participants With Significant Nausea
Description: Nausea (defined as the desire to vomit without the presence of expulsive muscular movements) measured on a 0-10 verbal response scale, where 0=no nausea at all and 10=the worst nausea imaginable. "Significant nausea" means a score ≥ 4.
Time Frame: 24 hours after end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | APD421 5mg + Standard Anti-emetic | Placebo + Standard Anti-emetic
Number analyzed (Participants) | 572 | 575
Participants | 212 | 274
Statistical Analysis 1: Comparison: APD421 5mg + Standard Anti-emetic vs Placebo + Standard Anti-emetic; Test type: Superiority; p < 0.001, Chi-squared

6. Secondary Outcome: Time to First Violation of Criteria for PONV
Description: Criteria for PONV are any episode of emesis or use of rescue medication in the 24 hours after the end of surgery
Time Frame: 24 hours after end of surgery
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | APD421 5mg + Standard Anti-emetic | Placebo + Standard Anti-emetic
Number analyzed (Participants) | 572 | 575
minutes | NA [195.5 to NA] — Median value not available as <50% of participants met criteria for PONV. Upper bound of IQR not available as <75% of participants met criteria for PONV. | 821.0 [107.0 to NA] — Upper bound of IQR not available as <75% of participants met criteria for PONV.
Statistical Analysis 1: Comparison: APD421 5mg + Standard Anti-emetic vs Placebo + Standard Anti-emetic; Test type: Superiority; p < 0.001, Log Rank

ADVERSE EVENTS:
Time Frame: For the 7 day period after study drug administration
Arm/Group | APD421 + Standard Anti-emetic | Placebo + Standard Anti-emetic
All-Cause Mortality (participants affected / at risk) | 1/572 | 0/575
Serious Adverse Events (participants affected / at risk) | 14/572 | 14/575
Other Adverse Events (participants affected / at risk) | 111/572 | 120/575
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APD421 + Standard Anti-emetic (N=572) | Placebo + Standard Anti-emetic (N=575)
Post Procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Wound Secretion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Herpatic Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic Organ Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoerative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Post Operative wound infections (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infections (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Small intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APD421 + Standard Anti-emetic (N=572) | Placebo + Standard Anti-emetic (N=575)
Nausea (Gastrointestinal disorders) | 62 (62) | 70 (70)
Procedural Pain (Injury, poisoning and procedural complications) | 53 (53) | 58 (58)

LIMITATIONS AND CAVEATS:
There were no limitations and caveats that occurred during the duration of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days